CLINICAL TRIAL: NCT05113836
Title: LIPId Profile Changes in Inflammatory Conditions Induced by SARS-CORoronavirus-2 : LIPICOR Study
Brief Title: LIPId Profile Changes in Inflammatory Conditions Induced by SARS-CORoronavirus-2
Acronym: LIPICOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP20128; 2020-A02638-3 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2021-10-11; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-08

CONDITIONS: SARS-CoV2 Infection
Keywords: Infecious disease; Sars-CoV2; COVID-19; LDL; HDL; SAA; PON-1
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — On admission to the intensive care unit, a deep nasopharyngeal swab will be performed.
  A 5 ml tube of blood on EDTA medium will be taken at the same time as the blood ionogram for the treatment at D1, D3 and D7.
  During the research, the collection will be kept in the Biochemistry Laboratory of the Bichat Claude Bernard Hospital for a period of 2 years.
  At the end of the research, the samples will be kept and the aliquots necessary for the lipoprotein characterisation + genotyping experiments will be transferred to the Natinal Institute of Medical Reasearch U1188 laboratory.
  At the end of the research, the samples may be used for further analyses not foreseen in the protocol which may prove interesting in the context of the pathology according to the evolution of scientific knowledge, provided that the patient is not opposed to this, after having been informed, as indicated in the information/consent form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Any patient hospitalised in intensive care for a COVID-19 infection.: Any patient hospitalised in intensive care for a COVID-19 infection. The health emergency of this pandemic and the potential therapeutic action of HDL particles justify the choice of this population for study.
  Interventions: Biological: Deep nasopharyngeal swab; Biological: Blood sample at D1, D3 and D7

INTERVENTIONS:
Biological: Deep nasopharyngeal swab — On admission in ICU, a deep nasopharyngeal swab will be performed (15mL).
Biological: Blood sample at D1, D3 and D7 — Specific samples for research and lipid analysis will be performed at D1, D3 and D7:
  Assessments will be carried out on the same blood tube as the blood ionogram carried out as part of the usual management.
  This means a 5 ml tube of blood on EDTA medium will be taken at the same time as the blood ionogram for the treatment at D1, D3 and D7 (15mL in total).

SUMMARY:
In late 2019, a new coronavirus called severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) was identified as the cause of COVID-19 (COronaVIrus Disease-2019) in Hubei Province, China. COVID-19 has become a pandemic with approximately 4.1 million confirmed cases as of May 2020 resulting in 280,000 deaths worldwide. Between 5 and 20% of patients hospitalized with SARS-CoV-2 infection are admitted to the ICU with a mortality ranging from 25 to 60% depending on the series. At present, there is no effective targeted therapy against this viral infection.

High-density lipoproteins (HDL) are nanoparticles made up of apolipoproteins, mainly apoA1, associated with phospholipids whose main function is the reverse transport of cholesterol from peripheral tissues to the liver. This property gives HDL a major cardiovascular protective effect. In addition to this effect, studies have highlighted a number of properties such as anti-inflammatory, anti-apoptotic, anti-thrombotic and anti-oxidant effects of these particles. Furthermore, it has been shown that HDL is able to bind and neutralize bacterial lipopolysaccharides (LPS), promoting their elimination.

During bacterial sepsis, a rapid decrease in plasma HDL cholesterol (HDL-C) concentration has been demonstrated, but also an inverse correlation between mortality and HDL-C concentration. In addition to the quantitative decrease in HDL during sepsis, dysfunctions of these particles have been described, such as major differences in size, or a notable alteration in protein composition with, in particular, more pro-inflammatory proteins. In this context of both quantitative and qualitative alteration of HDL, authors have tested the efficacy of injection of either reconstituted HDL (apoA1 + phosphatidylcholines) or peptides structurally similar to ApoA1 in animal models of sepsis and have demonstrated a protective effect on morbidity and mortality, with in particular a decrease in the inflammatory state induced by sepsis.

Low-density lipoproteins (LDL) can also neutralize LPS and observational studies have shown a decrease in the concentration of LDL cholesterol (LDL-C) during sepsis. The authors also showed that low LDL-C was associated with a poor prognosis in patients with sepsis.

During COVID-19-induced sepsis, a few studies have demonstrated a decrease in lipoprotein (HDL and LDL) concentration. More specifically, some authors have found an association between low lipoprotein concentrations and increased disease severity. To the best of the knowledge of the investigators, no study has specifically investigated particulate dysfunction of lipoproteins and in particular HDL during severe COVID-19 infections. On the other hand, as it has been described that lipoproteins and particularly HDL can bind bacterial components (LPS or LTA) favoring their clearance, it can be envisaged that these particles can also bind SARS-CoV-2 components, and this, in a more or less strong way depending on the virus strain.

The preliminary results of the investigators show that in sepsis, serum amyloid A (SAA) protein tends to replace apolipoprotein A1, making HDL dysfunctional. In addition, paraoxonase-1, an antioxidant enzyme mainly carried by HDL, is almost absent or degraded in septic patients. The SAA/PON-1 ratio could allow to assess the severity of COVID-19 damage and to reinforce a possible therapeutic strategy based on the supplementation of severe patients with apolipoprotein A1 and PON-1 rich HDL nanoparticles.

Main objective: To evaluate the functionality of HDL as a prognostic marker of mortality in COVID-19 patients in ICU. To do so, a quantification of the SAA/PON-1 ratio at plasma level and on isolated lipoproteins will be performed by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patient hospitalized in surgical intensive care unit for COVID-19 infection.

Exclusion Criteria:

* Pregnant or breastfeeding women
* CHILD B or C cirrhotic patients
* Moribund patients with an estimated life expectancy of less than 48 hours on admission to the ICU
* Subject protected by law under guardianship or curatorship
* No affiliation to a social security system
* Absence of signed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient hospitalised in intensive care for a COVID-19 infection. The health emergency of this pandemic and the potential therapeutic action of HDL particles justify the choice of this population for study.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2020-12-19 (Actual); Primary Completion 2022-01-05 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Change of concentration of Serum Amyloid A (SAA, inflammation protein) and paroxonase-1 (PON-1, antioxidant enzyme) in plasma and lipoproteins. | Day 1 and Day 7.
  The primary endpoint will be the change of concentration of Serum Amyloid A (SAA, inflammation protein) and paroxonase-1 (PON-1, antioxidant enzyme) in plasma and lipoproteins. SAA and PON-1 will be quantified by ELISA directly in plasma and after isolating by ultracentrifugation lipoproteins (HDL and LDL) from Day 1 and Day 7.

SECONDARY OUTCOMES:
Assessment of structural dysfunctions by proteomic approaches to lipoproteins during severe COVID-19 infections. | Day 1, Day 3 and Day 7
  Assessment of structural dysfunctions by proteomic approaches to lipoproteins during severe COVID-19 infections.
Quantification of plasma HDL-C, LDL-C and triglyceride concentrations over time in patients hospitalized in ICU for severe COVID-19 infection. | Day 1, Day 3 and Day 7
  Quantification of plasma HDL-C, LDL-C and triglyceride concentrations over time in
Study of HDL and LDL particle size profiles using the Lipo-print® technique. | Day 1, Day 3 and Day 7
  Study of HDL and LDL particle size profiles using the Lipo-print® technique.
Comparison of pro- and anti-inflammatory cytokines levels, such as IL-1 beta, IL-6, TNF-alpha, IL-10 or IL-18, in patients according to their particle dysfunction data. | Day 1, Day 3 and Day 7
  Comparison of pro- and anti-inflammatory cytokines levels, such as IL-1 beta, IL-6, TNF-alpha, IL-10 or IL-18, in patients according to their particle dysfunction data.
Comparison of particle dysfunction data to markers of endothelial dysfunction. | Day 1, Day 3 and Day 7
  Comparison of particle dysfunction data to markers of endothelial dysfunction.
Comparison of lipid profiles to the genotype of COVID-19 strains. | Day 1, Day 3 and Day 7
  Comparison of lipid profiles to the genotype of COVID-19 strains.
Search for binding of viral proteins to lipoproteins. | Day 1, Day 3 and Day 7
  Search for binding of viral proteins to lipoproteins.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien TANAKA, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bichat, Paris, France

REFERENCES:
- [Derived] Andrei S, Meilhac O, De Tymowski C, Snauwaert A, Stern J, Robert T, Lortat-Jacob B, Atchade E, Kantor E, Begue F, Montravers P, Tanaka S. Relationship between high-density lipoprotein cholesterol (HDL-C) concentration and ventilator-associated pneumonia in ICU COVID-19 patients. Anaesth Crit Care Pain Med. 2025 Aug;44(4):101535. doi: 10.1016/j.accpm.2025.101535. Epub 2025 May 1. PMID 40318849